CLINICAL TRIAL: NCT00343486
Title: An Eight- Week Randomized, Double-Blind, Placebo-Controlled, Parallel Group Proof of Concept Study to Assess the Efficacy, Safety and Tolerability as Well as the Pharmacokinetic Profile of Oral Solabegron (GW427353) 125mg and 50mg Administered Twice Daily vs Placebo in Women With Overactive Bladder
Brief Title: Dose Ranging Study Of Solabegron Versus Placebo In Female Patients With Overactive Bladder Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3P104833; M06-1605.
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — solabegron

INTERVENTIONS:
Drug: Solabegron

SUMMARY:
This study will test the effectiveness and safety of two doses of solabegron against placebo in reducing the symptoms of overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Overactive bladder with symptoms of urgency with urge incontinence and frequency which may be associated with nocturia but without bladder pain.
* Body mass index in the range of = 19 kg/m2 to <35 kg/m2.

Exclusion Criteria:

* Pregnant
* Of childbearing potential or willing to use specific barrier methods outlined in the protocol.
* Grade III/IV pelvic organ prolapse with or without cystocele.
* History of interstitial cystitis or bladder related pain.
* Stress incontinence or mixed incontinence where stress incontinence is the predominant component based on prior history.
* History of pelvic prolapse repair (cystocele or rectocele) or urethral diverticulectomy within six months of screening.
* Urinary incontinence due to causes other then detrusor over activity (e.g., overflow incontinence).
* Nocturnal enuresis only.
* Urinary retention, or other evidence of poor detrusor function.
* Current or history of Urinary Tract Infection.
* Diabetes insipidus.
* History of myocardial infarction, unstable angina, or Congestive heart failure.
* Chronic severe constipation.
* History of prior anti-incontinence surgery.
* History of radiation cystitis or a history of pelvic irradiation.
* Electrostimulation, biofeedback, or bladder training therapy (behavioral therapy) during the previous month prior to screening, or the intention to initiate such therapies during the study. Pessaries and implants are also excluded.
* Received any investigational product within 30 days of enrollment into the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2006-05

PRIMARY OUTCOMES:
Percent reduction in the number of incontinence episodes per 24 hrs after 8 weeks of treatment

SECONDARY OUTCOMES:
Improvement overactive bladder symptoms per 24 hrs after 4 and 8 weeks of treatment. Improvement in health related Qol. Descriptive statistics of solabegron and it's primary metabolite.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (57):
- Argentina (6):
  - GSK Investigational Site, Av Córdoba 2424, Buenos Aires
  - GSK Investigational Site, Bahía Blanca, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
- Australia (5):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Caboolture, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Spring Hill, Victoria
- Finland (2):
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Tampere
- France (4):
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Genis-Laval
  - GSK Investigational Site, Suresnes
- Germany (10):
  - GSK Investigational Site, Hagenow, Brandenburg
  - GSK Investigational Site, Schwedt, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Dessau, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Riga, Latvia
- Netherlands (6):
  - GSK Investigational Site, Apeldoorn
  - GSK Investigational Site, Emmen
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Tilburg
  - GSK Investigational Site, Utrecht
- New Zealand (4):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Whangarei
- Poland (2):
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
- Slovenia (3):
  - GSK Investigational Site, Celje
  - GSK Investigational Site, Ljubljana
  - GSK Investigational Site, Slovenj Gradec
- South Africa (3):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Somerset West
- GSK Investigational Site, Seoul, South Korea
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Donostia / San Sebastian
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo (Pontevedra)
- Taiwan (3):
  - GSK Investigational Site, Hualien City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei